CLINICAL TRIAL: NCT02255162
Title: Safety and Feasibility of Lenalidomide in Combination With HLA-mismatched Stem-cell Microtransplantation as Post-remission Therapy in Patients With Acute Myeloid Leukemia (AML)
Brief Title: Lenalidomide in Combination With Microtransplantation as Post-remission Therapy in AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigators, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-265
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myelocytic Leukemia; Acute Myelogenous Leukemia; Acute Granulocytic Leukemia; Acute Non-Lymphocytic Leukemia
Keywords: Acute Myeloid Leukemia (AML); Acute Myelocytic Leukemia; Acute Myelogenous Leukemia; Acute Granulocytic Leukemia; Acute Non-Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lenalidomide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  Participants will receive the following:
  * Cytarabine-intravenous, fixed dosage, given 5 times during cycle
  * HLA-mismatched stem-cell microtransplantation
  * Lenalidomide-administered daily per cycle
  Interventions: Drug: Lenalidomide; Genetic: HLA-mismatched stem-cell Microtransplantation; Drug: Cytarabine

INTERVENTIONS:
Drug: Lenalidomide — Patients will receive lenalidomide starting on day 6 of each post-remission cycle, following conclusion of cytarabine post-remission therapy on days 1-5. Following count recovery in the third post-remission cycle, patients will then receive lenalidomide daily as a maintenance therapy.
  Other Names: •Revlimid®
Genetic: HLA-mismatched stem-cell Microtransplantation — Patient will receive HLA-mismatched stem cell microtransplant infusion on day 6 of each post-remission cycle, following conclusion of course of cytarabine in each cycle.
Drug: Cytarabine — Patients will receive cytarabine post-remission therapy for 3 cycles, on days 1-5 of each cycle.
  Other Names: Cytosar-U ®; 1-β-Arabinofuranosylcytosine; Arabinosylcytosine; Cytosine arabinoside; Ara-C

SUMMARY:
This research study is evaluating the safety and tolerability of the drug lenalidomide in combination with and following mismatched related donor microtransplantation in high risk AML patients in first remission. This study also aims to define the maximum tolerated dose (MTD) of lenalidomide given in this setting.

Microtransplantation seeks to give the participant donor cells in hopes that those cells can attack the underlying cancer. However, since the donor cells do not replace all of the host cells, it can hopefully avoid many of the serious risks involved with standard transplant, including graft-vs.-host disease (GVHD) - a complication where the donor cells attack the participant's normal body. Recent studies have suggested that lenalidomide can help aid donor cells to attack cancer when given after a stem cell transplant. This trial is trying to see if lenalidomide can help encourage the attack of leukemia cells by donor cells given as part of microtransplantation.

The FDA (the U.S. Food and Drug Administration) has approved lenalidomide but it has been approved for other uses such as in the treatment of other cancers including multiple myeloma and non-Hodgkin lymphoma. Although lenalidomide has been studied in patients with AML, it has not been approved by the FDA for standard use in AML. Lenalidomide is a compound made by the Celgene Corporation. It has properties which could demonstrate antitumor effects. The exact antitumor mechanism of action of lenalidomide is unknown.

DETAILED DESCRIPTION:
After the screening procedures confirm that the participant is eligible to participate in the research study. The participant will be given a study drug-dosing calendar.

The investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants, not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well they have tolerated their doses. Participants will receive the following:

* Cytarabine
* Microtransplantation
* Lenalidomide

ELIGIBILITY:
Inclusion Criteria:

* Recipient Inclusion Criteria
* Adults, aged 18 through 75 years of age, with pathologically confirmed acute myelogenous leukemia, in pathologically confirmed complete remission following anti-leukemic therapy.
* AST, ALT and Alkaline Phosphatase <5x Upper Limit normal (ULN), direct bilirubin < 2.0 mg/dl.
* Adequate renal function as defined by: calculated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault Formula) or serum Cr less than institution ULN (the elderly will often have < 60 GFR)
* ECOG performance status 0-2.
* Have a diagnosis of high-risk AML as established by a poor-risk karyotype, adverse risk by ELN criteria, a therapy-related AML, age ≥ 60 or with antecedent hematologic disorder
* LVEF must be equal to or greater than 40%, as measured by MUGA scan or echocardiogram
* Patients, or appropriate designee, must be able to provide informed consent.
* Must not have received systemic anti-neoplastic therapy, including radiotherapy within 14 days of study treatment.
* Female patients of childbearing age must have negative pregnancy test.
* Male subject agrees to use an acceptable method for contraception during the entire study treatment period and through 6 months after the last dose of lenalidomide.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. If needed, patients should be able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation.
* Donor Inclusion Criteria
* Haploidentical 1st-degree relative as defined by 3/6 or 4/6 HLA-matched at HLA -A, -B, or -DRB1 who is 18-70 years of age
* ECOG performance status 0 or 1
* Excellent health per conventional pre-donor history (medical and psychosocial evaluation)
* No positive testing for viral infection (HbsAg, HIV, HCV)
* Donor ability to understand and provide informed consent
* Meets standard institutional criteria for GCSF mobilized PBSC donation

Exclusion Criteria:

* Recipient Exclusion Criteria
* Diagnosis of acute promyelocytic leukemia
* Active refractory or relapsed acute leukemia
* Prior use of fludarabine, as this agent has been associated with higher subsequent rates of graft versus host disease
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study drug. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* A diagnosis of active hepatitis B or C as defined by detectable viral load assays in the blood
* Known hypersensitivity to thalidomide or lenalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking lenalidomide.
* Significant cardiac disease as determined by the investigator including:

  * Known or suspected cardiac amyloidosis
  * Congestive heart failure of Class III or IV of the NYHA classification
  * Uncontrolled angina, hypertension or arrhythmia
  * Myocardial infarction in past 6 months
  * Any uncontrolled or severe cardiovascular disease
  * Prior cerebrovascular event with persistent neurologic deficit
* Medical conditions that, in the investigator's opinion, would impose excessive risk to the subject.
* Equal to or greater than grade 2 ataxia, cranial or peripheral neuropathy.
* Systemic infection requiring IV antibiotic therapy within 7 days preceding the first dose of study drug, or other severe infection.
* Pregnant women are excluded from this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of lenalidomide after microtransplantation | Baseline, 42 Days

SECONDARY OUTCOMES:
Disease Free Survival | 1 year
Overall Survival | 1 Year
To assess immunomodulatory effects of this combination through measurement of T cell subsets by flow cytometric techniques and through microchimerism analysis at multiple points on study | 2 Years
To identify incidence and severity of acute and chronic graft versus host disease (GVHD). | 2 Years
To detect and categorize, according to severity, the cumulative incidences of toxicities | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Amir Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided